CLINICAL TRIAL: NCT01205139
Title: A Phase I, 2-panel, Open-label, Randomized, Cross-over Trial in Healthy Subjects to Investigate the Pharmacokinetic Interaction Between TMC435 and Antiretroviral Agents, TMC278 and Tenofovir Disoproxil Fumarate (TDF), at Steady State
Brief Title: TMC435-TiDP16-C114 - A Study in Healthy Volunteers Investigating the Pharmacokinetic Interaction Between TMC435 and the Antiretroviral Agents TMC278 and Tenofovir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR017392
Record Dates: First submitted 2010-09-16; First posted 2010-09-20 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Hepatitis C Virus
Keywords: TMC435-TiDP16-C114; TMC435-C114; TMC435; HCV; Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Simeprevir; Rilpivirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 001 (Experimental): TMC435 150 mg capsule once daily for 11 days
  Interventions: Drug: TMC435
- 002 (Experimental): TMC278 25 mg tablet once daily for 11 days
  Interventions: Drug: TMC278
- 003 (Experimental): TMC435 + TMC278 150 mg TMC435 capsule + 25 mg TMC278 tablet once daily for 11 days
  Interventions: Drug: TMC435 + TMC278
- 004 (Experimental): TMC435 150 mg capsule once daily for 7 days
  Interventions: Drug: TMC435
- 005 (Experimental): TDF 300 mg tablet once daily for 7 days
  Interventions: Drug: TDF
- 006 (Experimental): TMC435 + TDF 150 mg TMC435 capsule + 300 mg TDF tablet once daily for 7 days
  Interventions: Drug: TMC435 + TDF

INTERVENTIONS:
Drug: TMC435 — 150 mg capsule once daily for 7 days
  Arms: 004
Drug: TDF — 300 mg tablet once daily for 7 days
  Arms: 005
Drug: TMC435 + TDF — 150 mg TMC435 capsule + 300 mg TDF tablet, once daily for 7 days
  Arms: 006
Drug: TMC435 + TMC278 — 150 mg TMC435 capsule + 25 mg TMC278 tablet, once daily for 11 days
  Arms: 003
Drug: TMC278 — 25 mg tablet once daily for 11 days
  Arms: 002
Drug: TMC435 — 150 mg capsule once daily for 11 days
  Arms: 001

SUMMARY:
The purpose of this study is to investigate the effect of steady-state concentrations of TMC435 on the steady-state pharmacokinetics of TMC278 or Tenofovir , and vice versa. Steady state is a term which means that the drug has been given long enough so that the plasma concentrations will remain the same with each subsequent dose. TMC435 is being investigated for the treatment of chronic hepatitis C virus (HCV) infection. TMC278 and Tenofovir are two antiretroviral drugs for treatment of human deficiency virus (HIV) infection. Pharmacokinetics (pk) means how the drug is absorbed into the bloodstream, distributed in the body and eliminated from the body.

DETAILED DESCRIPTION:
TMC435 is being investigated for treatment of chronic HCV infection, in combination with Peg-IFN (pegylated interferon) and RBV (ribavirin). About 30% of all HIV infected patients are co-infected with HCV and need treatment for both infections. The results of this study will provide dosing recommendations for coadministration of TMC435 and TMC278 or Tenofovir in HCV-HCV co-infected patients. This is a Phase I, open-label (both participant and investigator know the name of the medication given at certain moment), randomized (sequence of treatment with study medications is assigned by chance), crossover trial in 48 healthy participants to investigate the pharmacokinetic interaction between TMC435 and an antiretroviral agent (TMC278 or tenofovir), at steady state. The participants are being allocated to one of two panels. In Panel 1, participants will receive three treatments (treatment A-B-C) in a randomized order. Participants will receive TMC435 150 mg q.d., TMC278 25 mg q.d.and TMC278 25 mg q.d. + TMC435 150 mg q.d., respectively. All treatments will be administered for 11 days and with food. There will be a washout period (a period where no study drug will be taken in view of having all the medication eliminated from the body before starting a new treatment) of at least 14 days between last intake of study medication in one session and first intake of study medication in the subsequent session. In Panel 2, participants will receive three treatments (treatment D-E-F) in a randomized order. Participants will receive TMC435 150 mg q.d., TDF 300 mg q.d. and TDF 300 mg q.d. + TMC435 150 mg q.d., respectively. All treatments will be administered for 7 days and with food. There will be a washout period of at least 7 days. Pharmacokinetic profiles of all three compounds will be determined through blood samples taken at regular intervals during the study. Safety and tolerability will be assessed during the study period and in follow-up. Blood and urine samples, electrocardiogram (ECG) and vital signs (blood pressure and heart rate) will be taken at screening, before medication intake on days 1 and 11 and on Day 12 in each session of Panel 1, before medication intake on days 1 and 7 and on Day 8 in each session of Panel 2, 5 hours post dose on Day11 and Day 7 in Panel 1 and 2, respectively and at the 2 follow up visits at 1 week and 4-5 weeks after last dose of study medication in the last session. A physical examination will be performed at screening, on day -1 (= day before first medication intake in each session for both panels) and during the 2 follow up visits. Each volunteer will receive 3 treatments for 11 or 7 days (Panel 1 and 2, respectively), minimum 14 or 7 days apart from each other (Panel 1 and 2, respectively). Volunteers in Panel 1 will take oral TMC435 150 mg q.d., oral TMC278 25 mg q.d. and combined. Volunteers in Panel 2 will take oral TMC435 150 mg q.d., oral TDF 300 mg q.d. and combined.

ELIGIBILITY:
Inclusion Criteria:

* No-smoker for at least 3 months
* Body Mass Index of 18.0 to 30.0 kg/m2
* Healthy based on a medical evaluation including medical history, physical examination, blood tests and electrocardiogram

Exclusion Criteria:

* Infection with Hepatitis A, B or C Virus
* Infection with the Human Immunodeficiency Virus (HIV)
* History of, or any current medical condition which could impact the safety of the participant in the study
* Having previously participated in a multiple-dose trial with TMC435 and/or TMC278, or in a single- or multiple-dose trial with TMC278 long-acting
* Having previously participated in more than 3 single-dose trials with TMC435 and/or TMC278.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2010-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Rate and extent of absorption of TMC435 following co-administration with TMC278 under fed condition, and vice versa. | Measured on Day1, 9, 10, 11 and 12 per treatment in Panel 1.
Rate and extent of absorption of TMC435 following co-administration with TDF under fed condition, and vice versa. | Measured on Day1, 5, 6, 7 and 8 per treatment in Panel 2.

SECONDARY OUTCOMES:
Safety and tolerability following co-administration of TMC435 and TMC278 (Panel 1) | 89 to 94 days (till and including last safety follow-up visit) for Panel 1
Safety and tolerability following co-administration of TMC435 and TDF (Panel 2) | 63 to 68 days (till and including last safety follow-up visit) for Panel 2

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited